CLINICAL TRIAL: NCT01592396
Title: A Phase 1, Open-label Study to Evaluate the Pharmacokinetics of Tralokinumab in Adolescents With Asthma
Brief Title: A Phase 1, Open-label Study to Investigate the Pharmacokinetics of Tralokinumab (CAT-354) in Adolescents With Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-RI-CAT-354-1054; 2011-005503-33 (EudraCT Number)
Record Dates: First submitted 2012-04-25; First posted 2012-05-07 (Estimated); Results first posted 2017-01-20 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Asthma
Keywords: Tralokinumab; CAT-354; Asthma
MeSH Terms: conditions — Asthma | interventions — tralokinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tralokinumab 300 mg (Experimental): Participants aged 12 to 14 years and 15 to 17 years will receive a single dose of tralokinumab (CAT-354) 300 milligram (mg), subcutaneously on Day 1.
  Interventions: Biological: Tralokinumab 300 mg

INTERVENTIONS:
Biological: Tralokinumab 300 mg — Participants aged 12 to 14 years and 15 to 17 years will receive a single dose of tralokinumab (CAT-354) 300 mg, subcutaneously on Day 1.
  Other Names: CAT-354

SUMMARY:
The pharmacokinetic (PK) profile of tralokinumab (CAT-354) will be studied in adolescent subjects with asthma.

DETAILED DESCRIPTION:
Interleukin-13 (IL-13) is a pleiotropic cytokine that promotes inflammation, airways hyper-responsiveness (directly and through recruitment and activation of inflammatory cells), mucus hypersecretion, airway remodeling via fibrosis, increased immunoglobulin E (IgE) synthesis and mast cell activation.Tralokinumab (CAT-354) is a human immunoglobulin G4 (IgG4) anti-IL-13 monoclonal antibody that has been shown to potently and specifically neutralize IL-13 in preclinical models.This study will evaluate the PK profile of a single dose of tralokinumab administered subcutaneously at a dose of 300 mg in adolescent subjects with asthma to be compared with the PK data from completed studies in adults.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-17 years (inclusive)
* Weight greater than (>) 30 kilogram (kg)
* Asthma for a minimum of 6 months prior to Screening
* Effective birth control for both male and female participants in line with protocol details.
* Exclusion Criteria:
* Previously taken tralokinumab (the study drug)
* Employee of the clinical study site or any other individuals directly involved with the conduct of the study, or immediate family members of such individuals
* Pregnant or breastfeeding women
* Current smoker or cessation less than (<) 3 months prior to screening
* Known immune deficiency excluding asymptomatic selective immunoglobulin A
* History of cancer - Hepatitis B, C or human immunodeficiency virus (HIV) positive
* Any disease which may cause complications whilst taking the study drug.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2012-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Piper, MBBS, Study Director — MedImmune Ltd
Locations (3):
- Poland (3):
  - Research Site, Gliwice
  - Research Site, Karpacz
  - Research Site, Lodz

REFERENCES:
- [Background] Baverel PG, Jain M, Stelmach I, She D, Agoram B, Sandbach S, Piper E, Kuna P. Pharmacokinetics of tralokinumab in adolescents with asthma: implications for future dosing. Br J Clin Pharmacol. 2015 Dec;80(6):1337-49. doi: 10.1111/bcp.12725. Epub 2015 Oct 1. PMID 26182954
- See also: CD-RI-CAT-354-1054 Statistical Analysis Plan — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=165&filename=CAT354_1054_SAP_Aug14.pdf
- See also: CD-RI-CAT-354-1054 Redacted Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=165&filename=CAT354_CP1054_Protocol_Legal%20IP_Redacted_02Sep14.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 30 participants were screened, out of which 20 were randomized into the study. The reasons for screen failures were not meeting the inclusion/exclusion criteria, and/or consent withdrawal.
Groups:
- Tralokinumab 300 mg (Participants Aged 12-14 Years) - Cohort 1: Participants aged 12 to 14 years received a single dose of tralokinumab (CAT-354) 300 milligram (mg), subcutaneously on Day 1.
- Tralokinumab 300 mg (Participants Aged 15-17 Years) - Cohort 2: Participants aged 15 to 17 years received a single dose of tralokinumab (CAT-354) 300 mg, subcutaneously on Day 1.
Period: Overall Study
Arm/Group | Tralokinumab 300 mg (Participants Aged 12-14 Years) - Cohort 1 | Tralokinumab 300 mg (Participants Aged 15-17 Years) - Cohort 2
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Pharmacokinetic (PK) population included all participants who received the investigational product and had at least 1 detectable post dosing tralokinumab (CAT-354) serum concentration.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tralokinumab 300 mg (Participants Aged 12-14 Years) - Cohort 1 | Tralokinumab 300 mg (Participants Aged 15-17 Years) - Cohort 2 | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.6 (0.7) | 15.8 (0.9) | 14.2 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax)
Time Frame: 0 (predose), 3, 8 and 24 hours postdose on Day 1; Day 4, 6, 8, 10, 15, 22, 36 and 57
Population: as for baseline characteristics
Measure: Median (Full Range); unit: days
Groups:
- Tralokinumab 300mg (Participants Aged 15-17 Years) - Cohort 2: Participants aged 15 to 17 years received a single dose of tralokinumab (CAT-354) 300 mg, subcutaneously on Day 1.
Arm/Group | Tralokinumab 300 mg (Participants Aged 12-14 Years) - Cohort 1 | Tralokinumab 300mg (Participants Aged 15-17 Years) - Cohort 2
Number analyzed (Participants) | 10 | 10
days | 5.2 ((3.0-9.1)) [3.0 to 9.1] | 6.1 (2.9-9.0) [2.9 to 9.0]

2. Primary Outcome: Maximum Observed Serum Concentration (Cmax)
Time Frame: 0 (predose), 3, 8 and 24 hours postdose on Day 1; Day 4, 6, 8, 10, 15, 22, 36 and 57
Population: PK population included all participants who received the investigational product and had at least 1 detectable post dosing tralokinumab (CAT-354) serum concentration.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Tralokinumab 300 mg (Participants Aged 12-14 Years) - Cohort 1 | Tralokinumab 300mg (Participants Aged 15-17 Years) - Cohort 2
Number analyzed (Participants) | 10 | 10
microgram per milliliter (mcg/mL) | 57.0 (21.7) | 50.6 (16.2)

3. Primary Outcome: Area Under the Concentration-time Curve From Zero to Infinity (AUC [0-infinity])
Description: AUC (0 - infinity) = Area under the serum concentration versus time curve (AUC) from time zero (predose) to extrapolated infinite time (0 - infinity). It is obtained from AUC (0 - t) plus AUC (t - infinity).
Time Frame: 0 (predose), 3, 8 and 24 hours postdose on Day 1; Day 4, 6, 8, 10, 15, 22, 36 and 57
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: (microgram*day)/milliliter (mcg*day/mL)
Arm/Group | Tralokinumab 300 mg (Participants Aged 12-14 Years) - Cohort 1 | Tralokinumab 300mg (Participants Aged 15-17 Years) - Cohort 2
Number analyzed (Participants) | 10 | 10
(microgram*day)/milliliter (mcg*day/mL) | 1916.0 (806.3) | 1721.1 (568.5)

4. Primary Outcome: Area Under the Concentration-Time Curve From Zero to Last Measurable Concentration (AUC [0-t])
Time Frame: 0 (predose), 3, 8 and 24 hours postdose on Day 1; Day 4, 6, 8, 10, 15, 22, 36 and 57
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg*day/mL
Arm/Group | Tralokinumab 300 mg (Participants Aged 12-14 Years) - Cohort 1 | Tralokinumab 300mg (Participants Aged 15-17 Years) - Cohort 2
Number analyzed (Participants) | 10 | 10
mcg*day/mL | 1561.4 (614.9) | 1384.6 (421.6)

5. Primary Outcome: Terminal Phase Elimination Half Life (t1/2)
Description: Terminal phase elimination half-life is the time measured for the serum concentration to decrease by one half.
Time Frame: 0 (predose), 3, 8 and 24 hours postdose on Day 1; Day 4, 6, 8, 10, 15, 22, 36 and 57
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tralokinumab 300 mg (Participants Aged 12-14 Years) - Cohort 1 | Tralokinumab 300mg (Participants Aged 15-17 Years) - Cohort 2
Number analyzed (Participants) | 10 | 10
days | 21.4 (5.5) | 22.1 (3.5)

6. Secondary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between administration of study drug and up to Day 57 that were absent before treatment or that worsened relative to pre-treatment state. Adverse events were summarized together for all participants.
Time Frame: Day 1 to Day 57
Population: Safety population included all participants who received investigational product.
Measure: Number; unit: participants
Arm/Group | Tralokinumab 300 mg
Number analyzed (Participants) | 20
participants
  TEAEs | 6
  TESAEs | 0

7. Secondary Outcome: Number of Participants Exhibiting Anti-Drug Antibodies for Tralokinumab at Any Visit
Description: Immunogenicity assessment included determination of anti-drug antibodies to tralokinumab (CAT-354) antibodies in serum samples. Immunogenicity results were summarized together for all participants.
Time Frame: Day 1 and Day 57
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- Tralokinumab 300mg: Participants aged 12 to 14 years and 15 to 17 years will receive a single dose of tralokinumab (CAT-354) 300 mg, subcutaneously on Day 1.
Arm/Group | Tralokinumab 300mg
Number analyzed (Participants) | 20
participants | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Day 57
Description: Adverse events were summarized together for all participants.
Arm/Group | Tralokinumab 300 mg
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 6/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tralokinumab 300 mg (N=20)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Injection site pruritus (General disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (4)
Pharyngitis (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Dose-normalized AUC(0-infinity) and dose-normalized Cmax were not evaluated as they were not relevant for single-dose study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The Principal Investigator (PIs) also agree for data to be presented first as a joint, multi-center publication.